CLINICAL TRIAL: NCT05136794
Title: Opioid Free Anaesthesia in Cardiac Surgery With Cardiopulmonary Bypas
Brief Title: LIdocaine veRsus Sufentanil Anaesthesia in Cardiac Surgery With Cardiopulmonary Bypass
Acronym: LISRACC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GUINOT 2021-4
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Opioid Free Anaesthesia; Opioid Anaesthesia
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opioid free anaesthesia: patient anesthtesized with lidocaine
  Interventions: Other: Data collection
- Opioid anaesthesia: patients anesthetized with sufentanil
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — complications: cardiac, neurological, renal, respiratory, red blood transfusion Hospital stays: ICU stays and hospital stay

SUMMARY:
Since the 90's the concept of morphine sparing and morphine free anaesthesia (OFA) has progressively developed in non-cardiac surgery. The principle is based on the fact that in a sleeping patient a sympathetic reaction marked by hemodynamic modifications does not translate into a painful phenomenon, that a painful phenomenon in a sleeping patient is not memorized, that hormonal stress, the sympathetic reaction and the inflammatory reaction can be controlled by other therapeutic classes than a morphine agent. This therapeutic management would avoid the side effects associated with the use of morphine. In this hypothesis, OFA is more and more practiced in various situations without the real impact in terms of clinical benefit being clearly demonstrated. In cardiac surgery, some centers practice OFA with various protocols.The purpose of this work is to retrospectively evaluate over a defined period the incidence of postoperative complications, length of stay in the ICU/hospital, and death rate between patients managed with/without OFA based on lidocaine.

ELIGIBILITY:
Inclusion Criteria:

age over 18 years Cardiac surgery with cardiopulmonary bypass performed between January 2019 and June 2021

Exclusion Criteria:

LVAD Heart transplantation Incomplete data in relation to outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgical
Sampling Method: Non-Probability Sample
Enrollment: 1772 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
ICU stays (days) | Day 30
  Total stay in ICU in day

SECONDARY OUTCOMES:
Complications | Day 30
  cardiac, neurological, renal, respiratory, red blood transfusion
Hospital stays (days) | Day 30
  hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Guinot PG, Andrei S, Durand B, Martin A, Duclos V, Spitz A, Berthoud V, Constandache T, Grosjean S, Radhouani M, Anciaux JB, Nguyen M, Bouhemad B. Balanced Nonopioid General Anesthesia With Lidocaine Is Associated With Lower Postoperative Complications Compared With Balanced Opioid General Anesthesia With Sufentanil for Cardiac Surgery With Cardiopulmonary Bypass: A Propensity Matched Cohort Study. Anesth Analg. 2023 May 1;136(5):965-974. doi: 10.1213/ANE.0000000000006383. Epub 2023 Feb 10. PMID 36763521